CLINICAL TRIAL: NCT02030145
Title: Thoracic Lymphatic Pump Techniques for Reducing Lung Volumes in Persons With Chronic Obstructive Pulmonary Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated
Sponsor: A.T. Still University of Health Sciences (Other)
Collaborators: American Osteopathic Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AOA Grant #06-04-545; 06-04-545 (Other Grant/Funding Number: American Osteopathic Association)
Record Dates: First submitted 2011-07-22; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Pulmonary
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Classic Thoracic Lymphatic Pump (Active Comparator): Subjects begin with Classic Thoracic Lymphatic Pump, then crossover to Compressive Thoracic Lymphatic Pump after 4-week washout period.
  Interventions: Procedure: Compressive Thoracic Lymphatic Pump; Procedure: Classic Thoracic Lymphatic Pump
- Compressive Thoracic Lymphatic Pump (Experimental): Subjects begin with Compressive Thoracic Lymphatic Pump, then crossover to Classic Thoracic Lymphatic Pump after 4-week washout period.
  Interventions: Procedure: Compressive Thoracic Lymphatic Pump; Procedure: Classic Thoracic Lymphatic Pump

INTERVENTIONS:
Procedure: Compressive Thoracic Lymphatic Pump — This technique is a modification of the Classic Thoracic Lymphatic Pump where some pressure is maintained on the chest wall at the end of each exhalation and at the end of the third or fourth breathing cycle, during the inhalation phase, the hands are slowly removed from the chest wall, gradually releasing pressure on the chest without causing a sudden change in intrathoracic pressures.
  Other Names: Modified TLP
Procedure: Classic Thoracic Lymphatic Pump — This technique is well described in Chapter 68 of the Foundations for Osteopathic Medicine, 2nd Edition.
  Other Names: TLP

SUMMARY:
The primary goal of this line of research is to see if realistic manipulative protocols can be developed to produce sustained reductions in residual volume and improve pulmonary function parameters in people with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
This study is a prospective randomized crossover study to evaluate the effects of two different manipulation techniques on pulmonary function parameters in persons with COPD. Thirty-six (36) subjects will be enrolled in the study in order to complete the study with at least 30 subjects. Pulmonary function measures will include spirometry and lung volume. The pulmonary function testing will be done baseline, 30 minutes post-treatment, and 3 hours post-treatment. The study protocol treatment consists of a five-minute treatment session of one of the two studied treatment techniques given in a random order. After a washout period of at least four weeks, the subject will return for a second treatment session using the other technique.

ELIGIBILITY:
Inclusion Criteria:All subjects must be age 50 or older, have a history consistent with the diagnosis of COPD, and have documented airflow obstruction and an increased residual volume on pulmonary function testing. Airflow obstruction is defined as an FEV1/FVC ratio of 70 percent or less of the predicted value and a RV of 120 percent or greater of the predicted value.

-

Exclusion Criteria:Subjects will be excluded if they have received any form of manipulative treatment in the 3 months prior to enrolling in the study. Subjects with acute respiratory illness, such as an exacerbation of COPD, acute bronchitis, or pneumonia will be excluded from the study. Persons unable to cooperate and follow instructions to complete pulmonary function testing due to dementia or other cognitive disorders will be excluded as will persons with spinal scoliosis greater than 25 degrees, significant chest wall deformity, and acute rib or compression fracture of the vertebra, unstable angina, or unstable congestive heart failure.

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pulmonary function tests | 30 minutes and 3 hours post-treatment
  Tests will be conducted by body plethysmography utilizing the MedGraphics® 1085 Series™ to measure changes in pulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: Donald R. Noll, D.O., Principal Investigator — A.T. Still University of Health Sciences
Locations (1):
- A.T. Still University of Health Sciences, Kirksville, Missouri, United States